CLINICAL TRIAL: NCT00655551
Title: A Multicenter, Open-label Trial to Assess the Safety and Tolerability of a Single Intravenous Loading Dose of Lacosamide Followed by Oral Lacosamide Maintenance as Adjunctive Therapy in Subjects With Partial-onset Seizures
Brief Title: Safety of Intravenous Lacosamide Dose Followed by Twice Daily Oral Lacosamide in Subjects With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0925; 2014-004378-40 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2008-03-26; First posted 2008-04-10 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: Partial Epilepsies; Partial Onset Seizures
Keywords: epilepsy; seizures; Lacosamide; Vimpat; intravenous
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lacosamide 200 mg cohort (Experimental): Single loading dose of intravenous (iv) lacosamide 200 mg followed by 6.5 days of oral lacosamide 100 mg twice daily
  Interventions: Drug: lacosamide
- Lacosamide 300 mg combined cohorts (Experimental): Single loading dose of intravenous (iv) lacosamide 300 mg dose followed by 6.5 days of oral lacosamide 150 mg twice daily
  Interventions: Drug: lacosamide
- Lacosamide 400 mg cohort (Experimental): Single loading dose of intravenous (iv) lacosamide 400 mg followed by 6.5 days of oral lacosamide 200 mg twice daily
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — Single loading intravenous (iv) lacosamide 200 mg dose administered over a 15 minute infusion duration followed by oral lacosamide 200 mg/day (100 mg twice daily) for 6.5 days
  Other Names: Vimpat
  Arms: Lacosamide 200 mg cohort
Drug: lacosamide — Single loading intravenous (iv) lacosamide 300 mg dose administered over a 15 minute infusion duration followed by oral lacosamide 300 mg/day (150 mg twice daily) for 6.5 days
  Other Names: Vimpat
  Arms: Lacosamide 300 mg combined cohorts
Drug: lacosamide — Single loading intravenous (iv) lacosamide 400 mg dose administered over a 15 minute infusion duration followed by oral lacosamide 400 mg/day (200 mg twice daily) for 6.5 days
  Other Names: Vimpat
  Arms: Lacosamide 400 mg cohort

SUMMARY:
The purpose of the trial is to evaluate the safety of intravenous (iv) lacosamide delivered in a single dose followed by 6.5 days of oral lacosamide treatment in subjects with partial-onset seizures.

DETAILED DESCRIPTION:
This multicenter, open-label trial examined safety and tolerability of rapid initiation of adjunctive lacosamide via a single intravenous loading dose followed by oral maintenance treatment in subjects 16 - 60 years of age with partial-onset seizures. Three consecutive 25-subject cohorts were given a progressively increasing dose of lacosamide (200, 300, 400 mg) administered as a single 15-minute intravenous (iv) loading dose followed by the equivalent daily dose administered orally twice daily for 6.5 days with the first oral dose 12 hours after the iv dose. A fourth cohort of 25 subjects repeated the 300 mg dose to provide safety data on a total of 50 subjects at the highest well-tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy with simple partial seizures and/or complex partial seizures
* Stable dose regimen of 1 to 2 marketed antiepileptic drug(s) (AED(s)) for 28 days prior to screening and duration of trial
* Acceptable candidate for venipuncture and intravenous (iv) infusion
* At least 1 partial seizure with motor component per 90 days
* Maximum allowed seizure frequency during 28 days prior to screening is 40 partial seizures of any type

Exclusion Criteria:

* Previous use of lacosamide
* History of primary generalized seizures
* History of status epilepticus within last 12 months
* History of cluster seizures during 8 week period prior to screening
* Non-epileptic events, including psychogenic seizures that could be confused with seizures
* Use of neuroleptics, monoamine oxidase (MAO) inhibitors, barbiturates, or narcotic analgesics within 28 days prior to screening
* Received any rescue benzodiazepines more than once during the 28 days prior to screening
* Concomitant treatment of felbamate or previous felbamate therapy within last 6 months
* Prior or concomitant vigabatrin use

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (7):
- United States (7):
  - Phoenix, Arizona
  - Baltimore, Maryland
  - Chesterfield, Missouri
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Charlottesville, Virginia

REFERENCES:
- [Result] Fountain NB, Krauss G, Isojarvi J, Dilley D, Doty P, Rudd GD. Safety and tolerability of adjunctive lacosamide intravenous loading dose in lacosamide-naive patients with partial-onset seizures. Epilepsia. 2013 Jan;54(1):58-65. doi: 10.1111/j.1528-1167.2012.03543.x. Epub 2012 Jun 18. PMID 22708895
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Lacosamide (200 mg): Single loading dose of intravenous (iv) lacosamide 200 mg followed by 6.5 days of oral lacosamide 100 mg twice daily
- Lacosamide (300 mg): Single loading dose of intravenous (iv) lacosamide 300 mg dose followed by 6.5 days of oral lacosamide 150 mg twice daily
- Lacosamide (400 mg): Single loading dose of intravenous (iv) lacosamide 400 mg followed by 6.5 days of oral lacosamide 200 mg twice daily
Period: All Periods Combined
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Started | 25 | 50 | 25
Completed | 25 | 47 | 21
Not Completed | 0 | 3 | 4
Not completed — Adverse Event | 0 | 3 | 4
Period: Period 1 (up to 7 Days)
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Started | 25 | 0 | 0
Completed | 25 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2 (up to 7 Days)
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Started | 0 | 25 | 0
Completed | 0 | 24 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Period 3 (up to 7 Days)
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Started | 0 | 0 | 25
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 4
Period: Period 4 (up to 7 Days)
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Started | 0 | 25 | 0
Completed | 0 | 23 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg) | Total
Number analyzed (Participants) | 25 | 50 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 0 | 2
  Between 18 and 65 years | 25 | 48 | 25 | 98
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.77) | 38.6 (11.53) | 39.6 (12.24) | 39.0 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 26 | 9 | 49
  Male | 11 | 24 | 16 | 51
Region of Enrollment [Number; unit: participants]
  United States | 25 | 50 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During the Treatment Period (up to 7 Days)
Description: An Adverse Event (AE) is any untoward medical occurrence (eg, noxious or pathological changes) in a subject or clinical investigation subject compared with pre-existing conditions, that occurs during any period of a clinical trial including Pre-treatment, Run-In, Wash-Out, or Follow-Up Periods. An AE is defined as being independent of assumption of any causality (eg, to study or concomitant medication, primary or concomitant disease, or study design).
Time Frame: Treatment period (up to 7 days)
Measure: Number; unit: subjects
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Number analyzed (Participants) | 25 | 50 | 25
subjects | 17 | 42 | 20

2. Primary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event
Description: as for outcome 1
Time Frame: Entire trial period (up to 6 weeks), screening through safety follow-up period (2 weeks post last medication)
Measure: Number; unit: subjects
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Number analyzed (Participants) | 25 | 50 | 25
subjects | 0 | 3 | 4

3. Secondary Outcome: Number of Subjects With at Least One Adverse Event With an Onset Within 4 Hours of Start of Infusion
Description: as for outcome 1
Time Frame: 0-4 hours post start of the infusion
Measure: Number; unit: subjects
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Number analyzed (Participants) | 25 | 50 | 25
subjects | 5 | 24 | 16

ADVERSE EVENTS:
Time Frame: up to 7 days
Arm/Group | Lacosamide (200 mg) | Lacosamide (300 mg) | Lacosamide (400 mg)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/50 | 1/25
Other Adverse Events (participants affected / at risk) | 7/25 | 37/50 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (200 mg) (N=25) | Lacosamide (300 mg) (N=50) | Lacosamide (400 mg) (N=25)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (200 mg) (N=25) | Lacosamide (300 mg) (N=50) | Lacosamide (400 mg) (N=25)
Diplopia (Eye disorders) | 1 (1) | 3 (3) | 5 (6)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 8 (8) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 9 (9) | 3 (3)
Gait disturbance (General disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 23 (27) | 15 (19)
Somnolence (Nervous system disorders) | 0 (0) | 17 (18) | 9 (9)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4)
Paraesthesia (Nervous system disorders) | 2 (2) | 3 (3) | 1 (4)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Coordination abnormal (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.